CLINICAL TRIAL: NCT01042418
Title: Appetite Profile After Intake of Rye Breakfast Meal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swedish University of Agricultural Sciences (Other)
Collaborators: Lantmannen Research and Development (Unknown)
Responsible Party: Hanna Isaksson, Swedish University of Agricultural Sciences,
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: RPM537
Record Dates: First submitted 2010-01-04; First posted 2010-01-05 (Estimated); Last update posted 2010-01-05 (Estimated); Status verified 2010-01

CONDITIONS: Obesity Prevention
Keywords: satiety; grain structure; rye

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Whole kernel breakfast (Experimental)
  Interventions: Other: Effect of breakfasts with whole vs milled rye kernels on appetite
- Wheat reference breakfast (Placebo Comparator)
  Interventions: Other: Effect of breakfasts with whole vs milled rye kernels on appetite
- Milled kernel breakfast (Active Comparator)
  Interventions: Other: Effect of breakfasts with whole vs milled rye kernels on appetite

INTERVENTIONS:
Other: Effect of breakfasts with whole vs milled rye kernels on appetite — Iso-caloric portions of the three breakfast foods along with identical additional foods are tested in a cross over design

SUMMARY:
Food structure influence metabolic response including appetite. Whole grain foods include a wide range of products; cracked or cut kernels, rolled flakes or milled to flour and used in foods such as breads, breakfast cereals and pasta.

DETAILED DESCRIPTION:
The aim of the present study was to investigate if rye grain structure influence perceived appetite. A comparison of whole rye kernels and milled rye kernels were done in two study parts. In the first part the rye was served as porridge breakfasts and in the second one milled and whole kernels were included into bread breakfasts. In order to observe potential effects that would arise when the remains of the meal reaches the colon, the period of measurement was set to 8 h after intake of iso-caloric rye bread and rye porridge breakfasts.

A randomized, crossover design was used to compare the effects of iso-caloric breakfast meals on subjective appetite during 8 h after consumption.

ELIGIBILITY:
Inclusion Criteria:

* 20 and 60 years;
* body mass index (BMI) 18-27 kg/m2;
* habit of consuming breakfast, lunch and dinner every day
* willingness to comply with the study procedures

Exclusion Criteria:

* intake of medicine likely to affect appetite or food intake;
* any medical condition involving the gastrointestinal tract;
* eating disorder;
* smoking;
* consumption of more than three cups of coffee per day;
* change of body weight more than 10% three months prior to screening;
* consumption of any restricted diet such as vegan, gluten free, slimming etc.;
* pregnancy, lactation or wish to become pregnant during the study period

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2008-10; Primary Completion 2009-06 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Subjective appetite (hunger, satiety, desire to eat) | 8 hours

REFERENCES:
- [Derived] Isaksson H, Rakha A, Andersson R, Fredriksson H, Olsson J, Aman P. Rye kernel breakfast increases satiety in the afternoon - an effect of food structure. Nutr J. 2011 Apr 11;10:31. doi: 10.1186/1475-2891-10-31. PMID 21481225